# Post-exposure Prophylaxis or Preemptive Therapy for SARS-Coronavirus-2: A Pragmatic Randomized Clinical Trial

Short Title: COVID-19 PEP RCT

UMN IRB Number: STUDY00009267

**FDA IND:** 148257

ClinicalTrials.gov: NCT04308668

Principal Investigator: David R Boulware

**Draft or Version Number: 2.3** 

24 April 2020

#### CONFIDENTIAL

This document is confidential and the property of the University of Minnesota. No part of it may be transmitted, reproduced, published, or used by other persons without prior written authorization from the principal investigator.

#### STATEMENT OF COMPLIANCE

This protocol will utilize a single institutional review board (IRB) registered with the Office of Human Research Protections (OHRP) and issued a Federal Wide Assurance (FWA). The research will be reviewed and approved by the IRB and will be subject to continuing review [45 CFR 46.103(b)].

#### SIGNATURE PAGE

The signature below constitutes the approval of this protocol and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable US federal regulations and ICH guidelines.

| Site Investigator: | | | |
|--------------------|---------------|-------|-----------|
| Signed: | David Bouware | Date: | 4/24/2020 |
| | Name | = | |
| | Title | | |

| COVID-19 PEP RCT | Version 2.3 |
|------------------|---------------|
| | 24 April 2020 |

# TABLE OF CONTENTS

| | Pa | age | | |
|---|------|--------|-------------------------------------------|----|
| 1 | Key | y Rol | es | 1 |
| 2 | Bad | ckgro | ound Information and Scientific Rationale | 2 |
| | 2.1 | Bad | ckground Information | 2 |
| | 2.2 | Rat | ionale | 7 |
| | 2.3 | Pot | ential Risks and Benefits | 8 |
| | 2.3 | .1 | Potential Risks | 8 |
| | 2.3 | .2 | Known Potential Benefits | 9 |
| 3 | Obj | jectiv | res | 10 |
| | 3.1 | Stu | dy Objectives | 10 |
| | 3.2 | Stu | dy Outcome Measures | 10 |
| | 3.2 | .1 | Primary Outcome Measures | 10 |
| | 3.2 | .2 | Secondary Outcome Measures | 10 |
| 4 | Stu | idy D | esign | 11 |
| 4 | .1 [ | Desig | n | 11 |
| | 4.2 | Stu | dy participant duration | 12 |
| | 4.3 | Stu | dy procedures | 12 |
| | 4.4 | Ind | vidually identifiable health information: | 12 |
| | 4.5 | Sub | ostudies (if applicable) | 12 |
| 5 | Stu | dy E | nrollment and Withdrawal | 13 |
| | 5.1 | Sub | oject Inclusion Criteria | 13 |
| | 5.2 | Sub | oject Exclusion Criteria | 13 |
| | 5.3 | Tre | atment Assignment Procedures | 14 |
| | 5.3 | .1 | Randomization Procedures | 14 |
| | 5.3 | .2 | Reasons for Withdrawal | 15 |
| | 5.3 | .3 | Handling of Withdrawals | 15 |
| | 5.3 | .4 | Termination of Study | 15 |
| 6 | Stu | idy Ir | tervention/Investigational Product | 16 |
| | 6.1 | Stu | dy Product Description | 16 |
| | 6.1 | .1 | Acquisition | 16 |
| | 6.1 | .2 | Formulation, Packaging, and Labeling | 16 |

| С | OVID-1 | 9 PEP | | Version 2.3<br>4 April 2020 |
|---|---|---|---|---|
| | 6.1 | .3 | Drug Description: | 16 |
| | 6.1 | .6 | Product Storage and Stability | 18 |
| | 6.2 | Dos | sage, Preparation, and Administration of Investigational Product | 18 |
| | Dru | ıg/De | evice Handling: | 18 |
| | 6.3 | Mod | dification of Investigational Product for a Participant | 18 |
| | 6.4 | Acc | countability Procedures for the Investigational Product: | 18 |
| | 6.5 | Ass | sessment of Subject Compliance | 18 |
| | 6.6 | Cor | ncomitant Medications/Treatments | 18 |
| 7 | Stu | idy S | chedule | 19 |
| | 7.1 | Scr | eening | 20 |
| | 7.2 | Enr | rollment/Baseline | 20 |
| | 7.3 | Foll | low-up | 20 |
| | 7.4 | Fina | al Study Visit | 21 |
| | 7.5 | Ear | ly Termination Visit | 21 |
| | 7.6 | Uns | scheduled / Sick Visit | 21 |
| 8 | Stu | idy P | rocedures/Evaluations | 22 |
| | 8.1 | Clin | nical Evaluations | 22 |
| | 8.2 | Lab | oratory Evaluations | 22 |
| 9 | Ass | sessr | ment of Safety | 23 |
| | 9.1 | Spe | ecification of Safety Parameters | 23 |
| | 9.2 | Met | thods and Timing for Assessing, Recording, and Analyzing Safety Paramet | ters 23 |
| | 9.2 | .1 | Adverse Events | 23 |
| | 9.2 | .2 | Reactogenicity (for Vaccine Studies and Some Therapeutic Trials) | 23 |
| | 9.2 | .3 | Serious Adverse Events (SAEs) | 23 |
| | 9.2<br>Abr | | Procedures to be Followed in the Event of Abnormal Laboratory Test Valual Clinical Findings | ues or<br>23 |
| | 9.3 | Rep | porting Procedures | 23 |
| | 9.3 | .1 | Serious Adverse Events | 23 |
| | 9.3 | .2 | Regulatory Reporting | 24 |
| | 9.3 | .3 | Reporting of Pregnancy | 25 |
| | 9.4 | Тур | e and Duration of Follow-up of Subjects after Adverse Events | 25 |
| | 9.5 | Saf | ety Oversight (DSMB) | 25 |
| 1 | 0 0 | Clinica | al Monitoring | 26 |

| COVID-1 | 9 PEP RCT | Version 2.3 |
|---|---|---|
| 11 8 | Statistical Considerations | 24 April 2020<br><b>27</b> |
| 11.1 | Study Hypotheses | 27 |
| 11.2 | Sample Size Considerations | 27 |
| 11.3 | Planned Interim Analyses | 28 |
| 11.4 | Final Analysis Plan | 29 |
| 12 5 | Source Documents and Access to Source Data | 31 |
| 13 ( | Quality Control and Quality Assurance | 31 |
| 14 E | Ethics/Protection of Human Subjects | 32 |
| 14.1 | Ethical Standard | 32 |
| 14.2 | Institutional Review Board | 32 |
| 14.3 | Informed Consent Process | 32 |
| 14. | 3.1 Informed Consent/Assent Process (in Case of a Minor) | 32 |
| 14.4 | Exclusion of Women, Minorities, and Children | 33 |
| 14.5 | Subject Confidentiality | 33 |
| 14.6 | Future Use of Stored Specimens | 33 |
| 15 [ | Data Handling and Record Keeping | 34 |
| 15.1 | Data Management Responsibilities | 34 |
| 15.2 | Data Capture Methods | 34 |
| 15.3 | Types of Data | 34 |
| 15.4 | Timing/Reports | 34 |
| 15.5 | Study Records Retention | 34 |
| 15.6 | Protocol Deviations | 34 |
| 16 F | Publication Policy | 34 |
| 17 L | Literature References | 35 |

#### LIST OF ABBREVIATIONS

AE Adverse Event/Adverse Experience

CFR Code of Federal Regulations

CONSORT Consolidated Standards of Reporting Trials

CFR Code of Federal Regulations
COVID19 coronavirus disease 2019

SRS-CoV SARS coronavirus (i.e. circa 2003) SARS-CoV-2 SARS coronavirus 2 (i.e. circa 2019)

CRF Case Report Form

CRO Contract Research Organization
DCC Data Coordinating Center

DHHS Department of Health and Human Services

DMID Division of Microbiology and Infectious Diseases, NIAID, NIH

DSMB Data and Safety Monitoring Board eCRF Electronic Case Report Form FDA Food and Drug Administration

FWA Federalwide Assurance GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

ICF Informed Consent Form

ICH International Conference on Harmonisation

IDS Investigational Drug Services

IEC Independent or Institutional Ethics Committee

IND Investigational New Drug Application

IRB Institutional Review Board

MERS-CoV Middle East respiratory syndrome coronavirus

MOP Manual of Procedures

N Number (typically refers to subjects)

NIAID National Institute of Allergy and Infectious Diseases, NIH

NIH National Institutes of Health

OCRA Office of Clinical Research Affairs, DMID, NIAID, NIH, DHHS

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

ORA Office of Regulatory Affairs, DMID, NIAID, NIH, DHHS

PCR Polymerase chain reaction
PHI Protected Health Information

PI Principal Investigator
SAE Serious Adverse Event

SOP Standard Operating Procedure

US United States

WHO World Health Organization

## **Summary**

| Full Title: | Post-exposure prophylaxis or Preemptive Therapy for coronavirus: A Pragmatic Randomized Clinical Trial |
|---|---|
| Short Title: | COVID-19 PEP RCT |
| Clinical Phase: | III |
| Sponsor: | Investigator-Initiated Protocol, University of Minnesota |
| Principal Investigator: | David R Boulware, MD MPH |
| Accrual Ceiling | 3000 |
| Study Population | <ul> <li>Adult Household contacts or Healthcare workers exposed to persons with COVID-19 disease within 4 days (n=1500), or</li> <li>Non-hospitalized adults with symptomatic COVID-19 disease within 4 days of onset (n=1500)</li> </ul> |
| Objective | <ol> <li>Test if hydroxychloroquine can prevent development of<br/>COVID-19 disease after known exposure to the SARS-CoV2<br/>virus.</li> <li>Test if early preemptive therapy in non-hospitalized adults with<br/>symptomatic COVID-19 disease can prevent disease<br/>progression and hospitalization</li> </ol> |
| Study Design | Double-blind, randomized placebo-controlled clinical trial Internet-based trial driven by self-report. Study medicine delivered by FedEx to consented participants. Follow up through 14 days, with SAEs followed up to 90 days |
| Intervention Arm: | Hydroxychloroquine 200mg tablet. |

| 1 | 24 April 2 |
|---|---|
| | 800 mg orally once, followed in 6 to 8 hours by 600 mg, then 600 mg once a day for 4 consecutive days (5 days in total) |
| | (This is a modified malaria dosing for hydroxychloroquine) |
| Control Arm: | Placebo 4 tabs once, followed in 6 to 8 hours by 3 tabs, then 3 tabs once a day for 4 consecutive days (5 days in total) |
| Primary Endpoint in Asymptomatic Cohort | Incidence of COVID-19 disease within 14 days among those who are asymptomatic with known exposure |
| Primary Endpoint in Symptomatic Cohort | Change in symptom severity score (visual analog scale 0-10) over 14 days |
| Secondary Endpoints | <ol> <li>Incidence of Hospitalization for COVID-19 or death</li> <li>Incidence of confirmed SARS-CoV-2 detection</li> <li>Incidence of possible COVID-19 symptoms</li> <li>Incidence of all-cause study medicine discontinuation</li> <li>Severity of symptoms at Day 5 and 14 by visual analog scale</li> <li>Ordinal Scale of COVID-19 disease maximum severity at day 14 among those who are symptomatic at trial entry</li> </ol> |
| Duration of<br>Participation | <ul> <li>Recruitment and follow up will be internet-based.</li> <li>14 days of active participation</li> <li>Up to 90 days follow up for those with COVID-19 diagnosis to assess final outcome or dried blood spot collection for antibody serologies.</li> </ul> |
| Inclusion Criteria | <ul> <li>Exposure to COVID-19 within 4 days, either as: <ul> <li>Occupational exposure, or</li> <li>Household contact.</li> </ul> </li> <li>OR <ul> <li>Individual with symptomatic COVID-19 disease confirmed by PCR+ or by compatible symptoms with exposure to known PCR+ case with &lt;=4 days of symptoms.</li> </ul> </li> <li>Age &gt;=18 years of age <ul> <li>Provision of Informed Consent</li> </ul> </li> </ul> |
| Exclusion Criteria | <ul> <li>Current hospitalization</li> <li>Allergy to chloroquine or hydroxychloroquine</li> <li>Prior retinal eye disease</li> <li>Concurrent malignancy requiring chemotherapy</li> <li>Known Chronic Kidney disease, Stage 4 or 5 or dialysis.</li> </ul> |

| • | 24 April 2 |
|---|---|
| | <ul> <li>Known glucose-6 phosphate dehydrogenase (G6PD) deficiency.</li> <li>Known Porphyria</li> <li>Weight &lt;50 kg</li> <li>Structural or ischemic heart disease</li> <li>Personal or family history of QT prolongation</li> <li>Current use of: hydroxychloroquine, chloroquine, mefloquine, or cardiac medicines of: amiodarone, digoxin, dofetilide, flecainide, procainamide, propafenone, or sotalol</li> <li>Current use of QT prolonging medicines, including azithromycin (Refer to protocol for full list).</li> </ul> |
| Stratification | Randomization will be stratified by baseline status of COVID-19 disease vs. asymptomatic with exposure. Analyses will be separate for asymptomatic vs. symptomatic cohorts |
| Statistical<br>Assumptions | <ul> <li>10% attack rate for close contracts (or 10% progression of disease to hospitalization among those symptomatic at entry)</li> <li>Comparison of Proportions by Fisher's Exact test for disease incidence;</li> <li>Comparison of ordinal scale of disease severity by proportional odds model</li> <li>N=621 sample per arm has 90% power to detect a 50% relative risk reduction (i.e. ≤5.0%) in disease incidence or 50% decrease in the ordinal disease severity (to ≤4.25% disease incidence and ≤1% hospitalization).</li> <li>20% dropouts, inflates sample size to n=750 per arm</li> </ul> |

#### **Schematic of Study Design:**



If hospitalization occurs, this SAE will be followed for up to 90 days

For participants who develop symptomatic disease, they will be followed for up to 90 days to assess final outcome status in the event of hospitalization.

Stratification is based on symptom status at baseline

- 1. 1500 asymptomatic healthcare workers or household contacts exposed to COVID-19
- 2. 1500 symptomatic COVID-19 outpatients

## 1 KEY ROLES

#### Individuals:

Principal Investigator: David R. Boulware MD, MPH, CTropMed

Co-Investigator: Sarah Lofgren, MD

Co-Investigator: Alison Galdys, MD

Co-Investigator: Matthew Pullen, MD

Co-Investigator: Radha Rajasingham, MD

Co-Investigator: Caleb Skipper, MD

Medical Monitor: Mahsa Abassi, DO MPH

Pharmacologist: Melanie Nicol, PharmD, PhD

Biostatistician: Kathy H Hullsiek, PhD

Associate Statistician: Ananta Bangdiwala, MS

Associate Statistician: Nicole Engen, MS

**Institution:** Division of Infectious Diseases, Department of Medicine, University

of Minnesota, Minneapolis, MN

## 2 BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE

## 2.1 Background Information

#### Significance of Research Question/Purpose:

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a rapidly emerging viral infection causing COVID19. The current strategy uses a public health model of identifying infected cases, isolation, and quarantine to stop transmission. Once exposed, observation is standard-of-care.

No effective therapy currently exists for treatment. The lack of effective therapy diminishes persons presenting post-exposure for self-quarantine. Having an effective post-exposure prophylaxis, even if only partially effective, may additionally create synergy for the public health strategy of case identification and isolation – if a safe prophylaxis is available.

People who develop COVID-19 disease generally develop signs and symptoms, including mild respiratory symptoms and fever, after an average of 5-6 days after exposure (i.e. mean incubation period). The range of the incubation period is between 1 to 14 days.[1]

Most people infected with the COVID-19 virus have mild disease and recover. Approximately 80% of laboratory-confirmed patients have had mild to moderate disease, which includes non-pneumonia and pneumonia cases, 14% have severe disease, and 6% are critically ill with respiratory failure, shock, and/or multiple organ dysfunction [1].

#### Preliminary Data:

Chloroquine has *in vitro* activity in cell lines against SARS-CoV and SARS-CoV2. In a Vero E6 cell line, the half-maximal effective concentration (EC50) activity of chloroquine was 1.13 µM against SARS-CoV2 [2]. Hydroxychloroquine is functionally equivalent as chloroquine.

Another compound under treatment trials, remdesivir (Gilead) had an EC50 of 0.77  $\mu$ M [2]. Remdesivir (Gilead) is not FDA-approved and in limited quantities. Hydroxychloroquine is FDA-approved and globally is inexpensive. Chloroquine is no longer broadly available in the USA.

#### Existing Literature:

Several drugs, such as ribavirin, interferon, lopinavir-ritonavir, corticosteroids, have been used in patients with SARS or MERS, although the efficacy is poorly understood as a gold standard randomized clinical trial has not been conducted.

After the original 2003 SARS outbreak, screening of compounds was performed. The Special Pathogens Branch of the Division of Viral and Rickettsial Diseases at the Centers for Disease Control and Prevention (CDC) in Atlanta, Georgia investigated chloroquine.

CDC investigators reported that post-infection chloroquine treatment was effective in vitro at preventing the spread of SARS-CoV infection in an in vitro cell-based system [3]. Vincent et al reported:

"In order to investigate the antiviral properties of chloroguine on SARS-CoV after the initiation of infection, Vero E6 cells were infected with the virus and fresh medium supplemented with various concentrations of chloroquine was added immediately after virus adsorption. Infected cells were incubated for an additional 16–18 h, after which the presence of virus antigens was analyzed by indirect immunofluorescence analysis. When chloroguine was added after the initiation of infection, there was a dramatic dose-dependent decrease in the number of virus antigen-positive cells (Fig. 2A). As little as 0.1-1 µM chloroquine reduced the infection by 50% and up to 90-94% inhibition was observed with 33-100 µM concentrations (Fig. 2B). At concentrations of chloroquine in excess of 1 µM, only a small number of individual cells were initially infected, and the spread of the infection to adjacent cells was all but eliminated. A half-maximal inhibitory effect (EC50) was estimated to occur at  $4.4 \pm 1.0 \,\mu\text{M}$  chloroquine (Fig. 2C). These data clearly show that the addition of chloroquine can effectively reduce the establishment of infection and spread of SARS-CoV if the drug is added immediately following virus adsorption." [3]

Figure 2. Post-infection chloroquine treatment reduces SARS-CoV.





Vincent et al also reported: "Since we observed antiviral effects by chloroquine immediately after virus adsorption, we further extended the analysis by adding chloroquine 3 and 5 h after virus adsorption and examined for the presence of virus antigens after 20 h. We found that chloroquine was still significantly effective even when added 5 h after infection (Fig. 3); however, to obtain equivalent antiviral effect, a higher concentration of chloroquine was required if the drug was added 3 or 5 h after adsorption." [3]

Further experiments demonstrated that chloroquine impaired the terminal glycosylation of angiotensin-converting enzyme-2 (ACE2) receptor, which is the binding site for the envelope spike glycoprotein of SARS-CoV and SAR-CoV2 [3].

Conversely, chloroquine did <u>not</u> have activity against Middle East respiratory syndrome coronavirus (MERS-CoV), which may be related to MERS binding to CD26 receptor protein [4].

In a March 9, 2020 publication, hydroxychloroquine was found to have greater activity than chloroquine [5]. The SARS-CoV-2 EC 50 values for hydroxychloroquine were 6.14  $\mu$ M at 24 hours and 0.72  $\mu$ M at 48 hours, [5]. Conversely, chloroquine EC50 values were >100  $\mu$ M at 24 hours and 18.01  $\mu$ M at 48 hours [5]. This inhibition assay was performed with Vero cells using an infectious dose of 100 plaque forming units.

**Figure 3** displays the antiviral activities of hydroxychloroquine for treatment or prophylaxis against SARS-CoV-2 *in vitro* [5].





## **Existing Clinical Data**

There is accumulating clinical data on treatment of hospitalized patients with COVID-19 infection with chloroquine or hydroxychloroquine. These data have been summarized by Pastick et al. as of April 15, 2020 [6]. To date, there is no conclusive evidence of clinical benefit of hydroxychloroquine for treatment of hospitalized patients.

There have been no studies of early therapy or preventative therapy.

| Reference | Overall Findings | Limitations | Study<br>design | Number of patients | | Treatment regimen | Severity of illness<br>(As reported) | Location | Outcomes |
|---|---|---|---|---|---|---|---|---|---|
| | | | | HCQ | Control | | | | |
| | Hydroxychloroquine (HCQ) | | | | | | | | |
| Chen J, et al. [7] | No statistically significant differences in conversion rate by day 7 (86.7% vs. 93.3%, p>0.05). No difference in clinical outcomes between groups. | Full article only available in Chinese. Not peer-reviewed. Small sample size. | Randomize<br>d controlled<br>trial | 15 | 15 | 400mg HCQ for<br>5 days | Unknown severity;<br>patients had<br>symptoms for 6-7<br>days | Shanghai,<br>China | At two weeks, all patients had negative viral nucleic acid tests. |
| Gautret et<br>al. [8] | In unadjusted analyses, there were significantly reduced viral titers in the HCQ arm at day 6 (70% compared to 12.5% PCR negative, p<0.001). All six patients receiving HCQ and azithromycin were SARS-CoV-2 negative on day 6. | Study design. Small sample size/underpowered. Exclusion of six patients from analysis (no intention to treat analyses). Lack of long-term outcomes. | Non-<br>randomized<br>, non-<br>blinded,<br>open-label<br>trial | 26 | 16 | 600mg HCQ for<br>10 days | 17% were asymptomatic 61% had upper respiratory symptoms 22% had chest CT confirmed pneumonia | Marseille,<br>France | Six patients in the treatment arm were excluded from analysis (one died, three required ICU admission, one withdrew, one was lost-to-follow-up). |

| | 24 April 2020 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Chen Z, et<br>al. [9] | Time to clinical recovery and cough remission were shortened in the HCQ group; resolution of pneumonia was higher in the HCQ group (80.6% vs. 54.8%) Two HCQ patients had mild adverse reactions (rash, headache). | Small sample size. Not peer-reviewed. | Randomize<br>d, parallel-<br>group trial | 31 | 31 | 400mg HCQ for<br>5 days | Mild illness<br>(PaO2/FiO2 >300<br>mmHg) with chest<br>CT confirmed<br>pneumonia | Wuhan,<br>China | Four patients in the control group developed severe illness (not defined). |
| Molina et<br>al. [10] | 8/10 had positive nasopharyngeal swabs at days 5-6 (80%, 95% CI: 49-94). | Small sample size. Not peer-reviewed. | Prospective<br>open-label<br>study | 11 | 0 | 600mg HCQ for<br>10 days +<br>azithromycin<br>500mg x1, then<br>250mg | 10/11 were receiving supplemental O2 | Paris,<br>France | One patient died, two were transferred to the ICU, one had medications stopped secondary to QTc prolongation. |
| Gautret et<br>al. [11] | Reduced nasopharyngeal viral titers at day 7 (83% negative) and 8 (93%). Mean length of hospitalization of 5 days. | Study design. Small sample size. Short follow-up time. Not peer-reviewed. | Non-<br>randomized<br>, non-<br>blinded,<br>open-label<br>trial | 80 | 0 | 600mg HCQ for<br>10 days +<br>500mg,<br>followed by<br>250mg<br>azithromycin | 5% were<br>asymptomatic<br>54% had pneumonia<br>92% of patients had<br>a low national early<br>warning score<br>(NEWS) and mild<br>disease | Marseille,<br>France | Sixty-five (81.3%) patients survived to hospital discharge. Three patients required ICU admission and one died. |
| | Chloroquine (CQ) | | | | | | | | |
| Gao J et<br>al. [12] | CQ was stated to be superior to standard of care treatment in preventing exacerbation of pneumonia, reducing days to conversion rate, and shortening time to clinical recovery. | Combined patients from various ongoing studies. No statistical methodology. | Interim<br>report | 100 | 0 | Not reported,<br>likely varied<br>from trial to trial. | NA | Qingdao,<br>China | NA |

### 2.2 Rationale

Current standard of care is observation and quarantine after exposure to COVID19.

As of March 6, 2020, the CDC estimates that the transmission of SARS-CoV2 after a U.S. household close contract is 10.5% (95%Cl, 2.9 to 31.4%) [13]. Among all close contacts, the SARS-CoV2 transmission rate is estimated at 0.45% (95%Cl, 0.12 to 1.6%) by the CDC. These estimates are based on monitoring of travel-associated COVID19 cases. Conversely, in a setting with community transmission, the secondary attack rate in China was 35% (95%Cl, 27-44%) based on 48 transmissions among 137 persons in 9 index patients.

Chloroquine or Hydroxychloroquine may have antiviral effects against SARS-COV2 which may prevent COVID19 disease or early preemptive therapy may ameliorate disease severity. This trial will use a modification of standard malaria dosing of hydroxychloroquine to provide post-exposure prophylaxis / preemptive therapy.

Standard malaria treatment dosing is:

800mg once, then 400mg in 6-8 hours, then 400mg daily x 2 days (3 days in total).

We propose to dose for SARS-CoV-2 post-exposure prophylaxis at:

• 800mg once, then 600mg in 6-8 hours, then 600mg daily x 4 days (5 days in total).

The projected levels achieved will be approximately  $4.4~\mu\text{M}$  which is at or above the half maximal effective concentration (EC50) where 50% viral inhibition would occur. A delayed start to prophylaxis will be occurring -- based on the intrinsic delay from the exposure to case notification to trial enrollment, and to receipt of the first medication dose. Thereby, higher doses may be necessary as seen in the CDC study [3]. Thus a malaria loading dose sequence will be used, but with higher daily doses thereafter to target reaching the above the EC50.

As the incubation period is 2-14 days with a mean incubation period of 5-6 days, we seek to deliver post-exposure prophylaxis by the morning of day 4 at the latest. (<=3 days is an inclusion criteria). We recognize this may turn "post-exposure prophylaxis" into more of a "preemptive therapy" for some subjects who rapidly develop disease after trial randomization. If hydroxychloroquine does not prevent disease for some, preemptive therapy may ameliorate the COVID19 disease severity. Attenuated disease may in turn be associated with reduced rates of transmission.

#### 2.3 Potential Risks and Benefits

#### 2.3.1 Potential Risks

Short-term use of hydroxychloroquine is well-tolerated with a safe track record since 1955. The most common reported side effects include:

- headache, dizziness, ringing in your ears;
- nausea, vomiting, stomach pain;
- loss of appetite, weight loss;
- mood changes, feeling nervous or irritable;
- skin rash or itching; or
- hair loss.

GI side effects are minimized when taken with a meal or with milk. Antacid medications should be spaced apart by at least 4 hours.

Potential adverse effects by system, as listed on the FDA package insert:

- **Eye**: "Chloroquine retinopathy" is a rare side-effect of chronic use after multiple years of use. This has not occurred with <1 year of continuous use.
- Dermatologic Reactions: Bleaching of hair, alopecia, pruritus, skin and mucosal pigmentation, photosensitivity, and skin eruptions (urticarial, morbilliform, lichenoid, maculopapular, purpuric, erythema annulare centrifugum, Stevens-Johnson syndrome, acute generalized exanthematous pustulosis, and exfoliative dermatitis).
- Hematologic Reactions: Various blood dyscrasias such as aplastic anemia, agranulocytosis, leukopenia, anemia, thrombocytopenia (hemolysis in individuals with glucose-6-phosphate dehydrogenase (G-6-PD) deficiency).
- Gastrointestinal Reactions: anorexia, nausea, vomiting, diarrhea, and abdominal cramps. Isolated cases of abnormal liver function and fulminant hepatic failure.
- Cardiac Reactions: Long-term use (>1 year) has been associated with the development of cardiomyopathy and arrhythmias. Specifically, chronic use has been associated with a mean +25msec prolongation of the QT interval after a median use of 3.5 years in patients with autoimmune diseases. In a 2018 review of short term antimalarial treatment trials (n=1076 with chloroquine), no serious cardiac adverse events were reported among 35,548 participants [14]
- Allergic Reactions: Urticaria, angioedema, and bronchospasm have been reported
- Central Nervous System Reactions: Irritability, nervousness, emotional changes, nightmares, psychosis, headache, dizziness, vertigo, tinnitus, nystagmus, nerve deafness, convulsions, ataxia
- Miscellaneous Reactions: Weight loss, lassitude, exacerbation or precipitation of porphyria and non-light-sensitive psoriasis. Possible Hypoglycemia in persons with diabetes

#### On 24 April 2020, FDA issued a caution:

# FDA cautions against use of hydroxychloroquine or chloroquine for COVID-19 outside of the hospital setting or a clinical trial due to risk of heart rhythm problems

Close supervision is strongly recommended

"The FDA is aware of reports of serious heart rhythm problems in patients with COVID-19 treated with hydroxychloroquine or chloroquine, often in combination with azithromycin and other QT prolonging medicines. We are also aware of increased use of these medicines through outpatient prescriptions. Therefore, we would like to remind health care professionals and patients of the known risks associated with both hydroxychloroquine and chloroquine. We will continue to investigate risks associated with the use of hydroxychloroquine and chloroquine for COVID-19 and communicate publicly when we have more information."

"Hydroxychloroquine and chloroquine can cause abnormal heart rhythms such as QT interval prolongation and a dangerously rapid heart rate called ventricular tachycardia. These risks may increase when these medicines are combined with other medicines known to prolong the QT interval, including the antibiotic azithromycin, which is also being used in some COVID-19 patients without FDA approval for this condition. Patients who also have other health issues such as heart and kidney disease are likely to be at increased risk of these heart problems when receiving these medicines."

**Mitigation of Risk:** The inclusion / exclusion criteria exclude cardiac risk factors, chronic kidney disease, and anti-arrhythmia medicines. On 24 April, additional QT prolonging medicines are excluded.

#### 2.3.2 Known Potential Benefits

- There are no known benefits in humans for preemptive treatment.
- In vitro antiviral activity against SARS-CoV and SARS-CoV2 viruses.
- Chloroquine and Hydroxychloroquine have a long history of safe, effective use as an antimalarial, both acutely and long-term use.
- Chloroquine is being used therapeutically for severe COVID-19 disease in China and Korea.
- Commonly used as a chronic medication for autoimmune disorders (rheumatoid arthritis, systemic lupus erythematosus).
- Recent studies have shown potential broad antiviral effects in vitro at dosages below currently recommended clinical dosing, reducing risk of potential adverse effects listed above.

## 3 OBJECTIVES

## 3.1 Study Objectives

To determine if hydroxychloroquine is effective at prevention of COVID-19 disease or reducing disease severity.

## 3.2 Study Outcome Measures

#### 3.2.1 Primary Outcome Measures

#### Asymptomatic Cohort

 Incidence of COVID-19 disease within 14 days (among those asymptomatic at baseline)

#### **Symptomatic Cohort**

Change in symptom severity score (visual analog scale 0-10) over 14 days

#### 3.2.2 Secondary Outcome Measures

- Incidence of hospitalization or death
- Incidence of confirmed SARS-CoV-2 detection
- Incidence of symptoms compatible with COVID-19 (possible disease)
- Incidence of all-cause study medicine discontinuation or withdrawal
- Incidence of adverse reactions
- Symptom severity on day 5 or 14 via visual analog scale
- Ordinal Scale of COVID-19 Disease Severity at day 14 (among those who are symptomatic at trial entry)

Illness without hospitalization

Hospitalization (or post-hospital discharge)

Hospitalization with ICU stay or Death

Assessment of outcome measures will be primarily by self-report. As necessary, COVID19 disease will be verified from public health records, medical records, or death certificates. The primary endpoints are different for the two cohorts (those who are asymptomatic with known exposure; or those who are symptomatic at trial entry), and analyses will be done separately for the two cohorts.

The primary analysis will use PCR+ confirmed disease. However if the absence of sufficient testing supplies continues then outpatients will not be offered SARS-CoV-2 testing unless they are sick enough to be hospitalized. In that case an alternate a priori planned analysis will define incident COVID19 disease as a composite of SARS-CoV-2 PCR+ confirmed result OR symptomatic disease (i.e. possible) COVID-19 in those without testing.

## 4 STUDY DESIGN



If hospitalization occurs, this SAE will be followed for up to 90 days

There are two strata: 1) asymptomatic healthcare workers or household contacts exposed to COVID-19 (n=1500); 2) symptomatic COVID-19 disease (n=1500). Follow up will occur up to 90 days for those with symptomatic COVID-19 disease who become hospitalized.

## 4.1 DESIGN

Randomized, double-blind, placebo-controlled clinical trial, parallel design

- Intervention Arm: Hydroxychloroquine 800 mg orally once (4 tablets), followed in 6 to 8 hours by 600 mg (3 tabelts), then 600 mg once a day for 4 consecutive days (5 days in total)
- Control Arm: Vitamin Placebo 4 tablets orally once, followed in 6 to 8 hours by 3 tablets, then 3 tablets once a day for 4 consecutive days (5 days in total)

# 4.2 Study participant duration

- 14 days consisting of internet-based virtual visits
- For participants ill with COVID-19 disease who are hospitalized (an SAE), observational follow up will extend to up to 90 days to assess final outcome status of their SAE.
- Pregnant women have their fetal outcome assessed postpartum to exclude a teratogenic SAE.

## 4.3 Study procedures

- All procedures will consist of internet-based questionnaires completed by self-report.
- Informed consent is provided to access medical records to verify information, as necessary.
- Optional: blood spot will be collected at approximately day 14.
- Optional: daily cardiac monitoring with remote EKG reads of QTc interval.

## 4.4 Individually identifiable health information:

Name, date of birth, addresses, and phone number will be collected so as to prescribe study medication. Email addresses will be collected for communication. If participants are hospitalized, the hospitalization date will be collected.

# 4.5 Substudies (if applicable)

Additional sub-studies will undergo separate IRB approval, and these studies will involve separate informed consent. Consented participants will be queried as to if they wish to participate in future research.

- 1) Serology for Coronavirus Antibodies: New Participants will be offer an optional participation in self-collection of dried blood spots in order to measure serologies for antibodies. Participants who have already been consented and entered the trial, will be approached for amendment of consent. The purpose of serology testing is two-fold: First, to verify infection. Second, the prevalence of antibodies will be compared among symptomatic and asymptomatic persons with a scientific question of how many asymptomatic persons seroconvert after a high risk exposure in the absence of symptomatic illness. The exact serology methodology to be conducted will be determined, based on availability and diagnostic performance. Blood spot collection materials (e.g. 18g lancet, filter paper, bandaid, instructions, and return envelope). (Optional)
- Cardiac Monitoring with handheld EKG to check cardiac QTc interval once daily for the first 7 days as a safety substudy. (Optional)

## 5 STUDY ENROLLMENT AND WITHDRAWAL

Participants will undergo screening via internet-based forms. The screening and inclusion criteria will be based on self-report.

## 5.1 Subject Inclusion Criteria

- Exposure to a COVID19 case within <=4 calendar days as either:
  - Occupational exposure (healthcare worker, first responder, etc.)
  - Household contact

OR

- Symptomatic COVID-19 disease
  - Confirmed diagnosis with PCR+ SARS-CoV-2 within <=4 days of symptom onset</li>
     OR
  - Individual with compatible symptoms with exposure to known PCR+ SARS-CoV-2 case within 14 days AND compatible symptoms of fever, cough, or shortness of breath (and no available /pending testing for the individual)\*
- >= 18 years of age
- Provision of informed consent

## 5.2 Subject Exclusion Criteria

- Current Hospitalization
- Contraindication or allergy to hydroxychloroguine
- Retinal eye disease
- Concurrent malignancy requiring chemotherapy
- Known glucose-6 phosphate dehydrogenase (G-6-PD) deficiency
- Known chronic kidney disease, stage 4 or 5 or receiving dialysis
- Known Porphyria
- Weight < 50 kg
- Structural or ischemic heart disease
- Personal or Family history of prolonged QT
- Current use of: hydroxychloroquine, chloroquine, or cardiac medicines of: flecainide, Tambocor; amiodarone, Cordarone, Pacerone; digoxin or Digox, Digitek, Lanoxin; procainamide or Procan, Procanbid, propafenone, Rythmal; or sotalol.
- Current use of QT prolonging medicines of:
  - Antimicrobials: levofloxacin, ciprofloxacin, moxifloxacin, azithromycin, clarithromycin, erythromycin, ketoconazole, itraconazole, or mefloquine
  - Antidepressants: amitriptyline, citalopram, desipramine, escitalopram, imipramine, doxepin, fluoxetine, wellbutrin, or venlafaxine
  - Antipsychotic or mood stabilizers: haloperidol, droperidol, lithium, quetiapine, thioridazine, ziprasidone
  - Methadone
  - Sumatriptan, zolmitriptan

#### Rationale for inclusion / exclusion criteria:

\* As of 20 March 2020, testing is limited in many U.S. states and locales due to insufficient supplies. Thus, outpatient testing may not be available. A person with known exposure to a confirmed COVID-19 case with subsequent compatible symptoms is eligible for enrollment, if testing is not available. If a symptomatic person tests negative for SARS-CoV-2, they are <u>not</u> eligible for enrollment.

Mean Incubation period is ~5.2 days, thus we wish to limit enrollment to those with a higher risk of progression and deliver study medicine in a time period to intervene to prevent disease or ameliorate disease (i.e. start of study medicine by <=4 days after exposure). The current (as of March 17, 2020) delays in testing makes this window particularly tight, and it may need to be relaxed in the future via protocol amendment.

In clinical practice of tropical medicine, chloroquine or hydroxychloroquine are prescribed without any baseline laboratory testing or monitoring.

Chronic use of hydroxychloroquine for >1 year can cause retinopathy or cardiomyopathy, thus persons with baseline conditions will be excluded. Study medicine is excreted via the kidney with dose reduction recommended in CrCl <30 cc/min (Stage 4 Kidney Disease). G-6-PD deficiency is listed as a caution on the FDA label. G-6-PD testing is not routinely performed in clinical care prior to giving hydroxychloroquine prescriptions (unlike with primaquine). Medication exclusions are for possible drug-drug interactions, particularly with cardiac arrhythmia medicines with a caution on the FDA-package insert.

On April 20, 2020, FDA mandated exclusion of structural or ischemic heart disease; or personal or family history of prolonged QT.

On April 24, 2020, FDA issued a caution for QT prolongation in persons with heart disease, chronic kidney disease, or taking other QT prolonging medicines.

# 5.3 Treatment Assignment Procedures

#### 5.3.1 Randomization Procedures

Participants will be randomized via permuted block randomization. Randomization will be recorded on an electronic log by the pharmacy. Study investigators and subjects will be blinded. There will be separate randomization schedules for the two cohorts (asymptomatic with exposure or symptomatic).

#### **Masking Procedures**

Participants will be provided masked study medicine, shipped by courier (e.g. FedEx). The intervention vs. placebo will not be identical; however, participants and outcome assessors will be masked to their assignment.

#### 5.3.2 Reasons for Withdrawal

Participants may withdraw at any time point at their discretion.

### 5.3.3 Handling of Withdrawals

Withdraws will be counted as failures for the secondary endpoint of completion of study medication.

Participants who discontinue study medication will still be asked to complete the follow up visit schedule.

#### **5.3.4 Termination of Study**

This study may be prematurely terminated if there is sufficient reasonable cause, including but not limited to:

- Unexpected, significant, or unacceptable risk to subjects
- Interim analyses by the DSMB.
- Insufficient compliance with protocol requirements
- Data are not sufficiently complete and/or not evaluable
- Regulatory authorities decide that study should be terminated

If the study is prematurely terminated for harm, current subjects will complete follow up, and no further subjects will be enrolled. If the study is terminated due to benefit, then the study will immediately convert into an open-label prospective cohort to collect further observational data on the safety and efficacy of the intervention, up to the IRB approved recruitment limit.

# 6 STUDY INTERVENTION/INVESTIGATIONAL PRODUCT

# **6.1 Study Product Description**

## 6.1.1 Acquisition

FDA-approved formulation of hydroxychloroquine will be purchased.

## 6.1.2 Formulation, Packaging, and Labeling

The study medicines will be packaged by the MHealth Investigational Drug Services. Dispensed medications will be delivered by courier (e.g. Fedex) to study participants.

HN

Labels will include: "Caution: New Drug – Limited by Federal Law to investigational use. Keep out of reach of children."

## **6.1.3 Drug Description:**

Hydroxychloroquine sulfate

**6.1.4** Formulation: 200mg tablet ( = 155 mg base of chloroquine)

#### **6.1.5** Pharmacokinetics:

- Absorption: Rapid and almost completely
- Distribution: Widely distributed into body tissues
- Metabolism: Partially hepatic to main metabolyte of desethylchloroquine
- Excretion: Urine (>=50% as unchanged drug); acidification of urine increases elimination
- $C_{max} = 1.2 \text{ nmol/mL} = 1.2 \mu \text{mol/L} = 1.2 \mu \text{M}$  at 400mg single dose.[15]
- $T_{max} = 2.4 \text{ hours}$
- $T_{1/2} = 172 + 39 \text{ hours} = 7.1 + 1.6 \text{ days}$
- AUC<sub>last</sub> = 75.4 + 47 nmol/h/mL
- This C<sub>max</sub> is in the therapeutic window for SARS-COV2 activity.
- Steady state doses for 400mg dose is 974  $\mu$ g/L = 2.24  $\mu$ M [16], thus a 600mg dose should generate approximately 3.4  $\mu$ M, which is above the EC50 of viral inhibition of 1.3  $\mu$ M (EC50 = 50% inhibition; however, the more inhibition the better, likely).

#### Population PK parameter modeling: 5 day regimen



Figure courtesy of Dr. Mahmoud Al-Kofahi of College of Pharmacy, Univ. of Minnesota

The EC50 has been reported as 0.72  $\mu$ M [5], although this is not a precise measurement, and should be view with a range of error present (but not reported). The EC50 is the point of 50% maximal inhibition, so more drug would be better (balanced against toxicity and drug supply). The percentage of persons achieving a 24 hour level above the EC50 is as follows (**Figure**).



## 6.1.6 Product Storage and Stability

Store at room up to 30° C (86° F). Dispense in a tight, light-resistant container.

# 6.2 Dosage, Preparation, and Administration of Investigational Product

### **Drug/Device Handling:**

Hydroxychloroquine or placebo will be dispensed by the MHealth Investigational Drug Service (IDS) Pharmacy. To do so, study investigators will send a prescription to the IDS Pharmacy, the pharmacy will randomize the subject, and dispense the appropriate study medicine. The medicine will then be provided to research volunteers via FedEx / courier delivery in the United States.

## 6.3 Modification of Investigational Product for a Participant

With mild side effects, participants will be instructed to split the 3 tablet daily dosing into multiple times per day.

In the event of substantial side effects, participants may discontinue the study medication and stay in the study to complete follow up.

# 6.4 Accountability Procedures for the Investigational Product:

Accountability will be via self-report at the day 5 virtual visit.

# 6.5 Assessment of Subject Compliance

Adherence will be via self-report at day 5 virtual visit.

#### 6.6 Concomitant Medications/Treatments

Participants may receive other concomitant medications or therapies, and will be asked to report these in regards to other therapies received on day 1, day 14, and in the event of hospitalization.

## 7 STUDY SCHEDULE

# **Screening Online Questionnaire**

- Email <u>covid19@umn.edu</u> or go to <u>www.covidpep.umn.edu</u> if you have been exposed to or diagnosed with COVID19
- You will be sent an email with information about our clinical trial
- A URL link will be provided for you to take the online screening survey

## **Medication Shipped**

- Study medicine will be shipped overnight to your address
- Study medicine should arrive by 10:30am (Mon-Sat)
  - If you enroll after ~12pm on Sat or Sun, will arrive Tue.
- Take 4 tablets of the study medicine with some food or milk

# Online Survey (Day 1)

- You will receive an email with a link to an online survey from covidfaq@umn.edu. If not received, check your spam folder.
- Take the second dose of 3 tablets 6-8 hours after the first.
- Take other medicines >= 4 hours apart from the study medicine

# Study Days 2-4

- · You should take 3 tablets each morning
- If you develop upset stomach, you may separate the pills; for example 1 at breakfast, 1 at lunch, and 1 at dinner.
- We will send a brief Day 3 survey

# **Online Survey (Day 5)**

- You will receive an email with a link to an online survey
- This should be the same day you finish the study medicine
- A brief follow up survey will also be sent on Day 10 to ask if you have any COVID19 symptoms

# **End of Study Survey (Day 14)**

- You will receive an email with a link to an online survey
- Unless you have developed symptoms, this marks the end of the study. We will ask if you wish to participate in future studies.
- If you were hospitalized or have pending tests, we will reach out to you every 2 weeks.

## 7.1 Screening

- Baseline screening for eligibility
- Informed consent by self-administered
- This will be performed via a web-based form. Eligibility criteria will be by self-report.

#### 7.2 Enrollment/Baseline

Randomization (Day 0)

- Participants will be randomized by a computer-generated algorithm using a permuted block randomization sequence.
- Randomization will be stratified by symptomatic vs. asymptomatic status at baseline.
- Investigational pharmacy will dispense the masked study medicine
- Study personnel will then FedEx study medicine to the participant
- Participant will be sent an email to expect medication to arrive by 10:30am

## 7.3 Follow-up

#### **Day 1 Virtual visit**

- Verify receipt of study medicine
- Clinical status check-in
  - Participant starts study medicine (4 tabs), then 3 tabs in 6-8 hours, then 3 tabs daily.
- Query for SARS-CoV-2 testing
- Query for symptom status (0-10 visual analog scale of symptom severity)
- Query for hospitalization or SAEs
- Query for medication-related side effects / AEs

#### **Day 3 Virtual visit**

- Query for symptom status (0-10 visual analog scale of symptom severity)
- Query for hospitalization or SAEs
- Query for medication-related side effects / AEs

#### Day 5 Virtual visit

- Query for symptom status (0-10 visual analog scale of symptom severity)
- Assessment of adherence by self-report
- Completion of study medicine, which has a ~7 day half-life
- Query for study medicine side effects since enrollment
- Query for SARS-CoV-2 testing
- Query for hospitalization or SAEs

#### Day 10 Virtual visit

- Query for symptom status (0-10 visual analog scale of symptom severity)
- Query for SARS-CoV-2 testing

- Query for SARS-CoV-2 testing
- Query for hospitalization or SAEs

## 7.4 Final Study Visit

- Day 14 Visit
  - Query for symptom status (0-10 visual analog scale of severity)
  - Query for study medicine side effects since enrollment
  - Query for SARS-CoV-2 testing
  - Query for hospitalization or SAEs
  - Query for pregnancy status
  - Final outcome assessment
  - Assess other medicines used during study period
  - Optional dried blood spot collection, return in pre-paid envelope.

If participations have a SAE prior to the final study visit (e.g. hospitalization), the final resolution of the event will be followed until resolution or up to 90 days. The hospitalization eCRF will be sent in 14 days interval to assess clinical outcome / resolution of the hospitalization. Pregnancies will be followed through delivery to assess for any teratogenic SAE.

## 7.5 Early Termination Visit

If participants develop new / worsening symptoms of coronavirus, they will be directed to their healthcare provider and/or local public health authority for clinical care. We will follow up of hospitalized patients for resolution of their SAE for up to 90 days to assess their final outcome. Participants will be sent the Hospitalization eCRF 14 days after hospitalization is reported with repeats in 14 day intervals until the participant is discharged from the hospital.

### 7.6 Unscheduled / Sick Visit

Subjects will be provided a central email contact: <a href="mailto:faq.covid19@gmail.com">faq.covid19@gmail.com</a> as a contact point for questions or concerns. This email will forward to an on-call study physician who will call the participant to resolve their concerns.

## 8 STUDY PROCEDURES/EVALUATIONS

#### 8.1 Clinical Evaluations

Clinical evaluations are by self-report.

# 8.2 Laboratory Evaluations

SARS-COV-2 positivity is by self-report. Informed consent asks for access to medical records.

Follow up PCR testing within 14 days is asked on followed questionnaires. Pending test results at 14 days or during hospitalization will be queried for final results with repeat survey sent at day 28.

Informed consent will request permission to contact local public health authorities or their medical provider in the event of lost to follow up or COVID19 disease.

There is no incentive to be dishonest, and we believe healthcare workers in particular will take their responsibilities seriously.

An optional dried blood spot collection will be offered at day 14. At time of informed consent, participants may opt into this collection. The dried blood spots will be used for future serology testing. Participants who opt into this testing will be mailed: i) instructions; ii) Whatman filter paper for dried blood spot collection; iii) one time use lancet; iv) return envelope.

Participants who have entered the trial prior to dried blood spot being offered and are <90 days from study entry will be contact with the option for dried blood spot testing of their antibody serology.

## 9 ASSESSMENT OF SAFETY

## 9.1 Specification of Safety Parameters

Hydroxychloroquine has a track record of safety since its FDA-approval in 1955. As an already, FDA-approved medicine, this trial is designed as a pragmatic trial in the setting of a public health emergency.

# 9.2 Methods and Timing for Assessing, Recording, and Analyzing Safety Parameters

#### 9.2.1 Adverse Events

Hydroxychloroquine has an excellent safety track record, being first FDA-approved in 1955. Adverse events will not be captured, unless they result in hospitalization. See Serious Adverse Events below.

Expected adverse events would include normal events within the general population as well COVID19-related disease events which may include need for hospitalization, pneumonia, respiratory failure, sepsis, and death.

## 9.2.2 Reactogenicity (for Vaccine Studies and Some Therapeutic Trials)

Not applicable

## 9.2.3 Serious Adverse Events (SAEs)

Hospitalization or death are protocol-defined endpoints.

SAEs (e.g. hospitalizations) will be followed for up to 90 days to assess final outcome.

# 9.2.4 Procedures to be Followed in the Event of Abnormal Laboratory Test Values or Abnormal Clinical Findings

Not applicable

# 9.3 Reporting Procedures

#### 9.3.1 Serious Adverse Events

An AE or suspected adverse reaction is considered a serious adverse event (SAE) if it results in any of the following outcomes:

- Death
- Life-threatening adverse event (as below)
- Hospitalization
- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
- Congenital anomaly/birth defect.
- Important medical events that may not result in death, but are life-threatening, or require hospitalizations may be considered serious when, based upon appropriate medical judgment they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

Life-threatening adverse events: An AE is considered "life-threatening" if, in the view of either the site principal investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death. For life threatening AEs, subjects would be recommended /expected to be hospitalized.

Based on the known safety track record of hydroxychloroquine, this pragmatic protocol will focus on death, life-threatening AEs, and hospitalizations. Incapacity / permanent disability is a possibility with COVID19, but this is not associated with hydroxychloroquine. In the event of incapacity, the subject would be expected to be hospitalized.

Hydroxychloroquine and chloroquine are not known to cause teratogenic events and are viewed as safe in pregnancy, especially with short term use. With this trial's sample size, this will not further delineate this risk. COVID19 disease may indeed be teratogenic. For women who are pregnant, we will ask to follow them through the end of their pregnancy, and they will be sent a follow up eCRF at 1 month post-partum based on their reported estimated date of delivery as provided at the day 14 study visit.

Thus, the hospitalization or death secondary endpoint will capture relevant SAEs. For those with ongoing hospitalization at the day 14 study visit, participants will be queried in 14 day intervals with the hospital eCRF to assess their final clinical outcome.

### 9.3.2 Regulatory Reporting

As hydroxychloroquine is an FDA-approved medicine being used at standard dosing, reporting to regulatory authorities will occur in summary format after each DSMB reports and at a frequency of at least annually.

Serious unexpected suspected adverse reactions (SUSARs) which are not expected with COVID-19 nor listed in the FDA package insert will be reported to the IRB. Those SUSARS which are deemed by an independent medical monitor to be related to the study medicine will be reported to the FDA and IRB.

## 9.3.3 Reporting of Pregnancy

Chloroquine and hydroxychloroquine are not known to be teratogenic. Chloroquine and hydroxychloroquine can accumulate in neonatal eyes. Conversely, the risk of severe COVID-19 infection is unknown, but likely is a heightened risk in pregnant women. The CDC states, "We do not have information on adverse pregnancy outcomes in pregnant women with COVID-19. Pregnancy loss, including miscarriage and stillbirth, has been observed in cases of infection with other related coronaviruses (SARS-CoV and MERS-CoV) during pregnancy. High fevers during the first trimester of pregnancy can increase the risk of certain birth defects."

Thus, the risk/benefit would favor the enrollment of women who may be or are pregnant, so as to not discriminate against pregnant women.

For women who are pregnant, we will ask to have follow through the end of their pregnancy to assess outcome of the pregnancy via a brief survey.

# 9.4 Type and Duration of Follow-up of Subjects after Adverse Events

Participants who are hospitalized for COVID-19 or SAEs will have up to 90 day follow up conducted to assess their final outcome. Management will be as per the participant's local healthcare provider.

# 9.5 Safety Oversight (DSMB)

A data and safety monitoring board (DSMB) will oversee the trial. The quorum will include three members and a biostatistician. The PI will be a non-voting observer, providing input as requested. See the DSMB charter for more details.

## 10 CLINICAL MONITORING

Clinical site monitoring is conducted to ensure that the rights and well-being of trial subjects are protected and that the reported trial data are accurate, complete, and verifiable. Clinical monitoring also ensures that conduct of the trial is in compliance with the currently approved protocol/ amendment(s), ICH, GCP, and with applicable regulatory requirement(s) and Sponsor requirements. Clinical monitoring will also verify that any critical study procedures are completed following specific instructions. Monitoring will be the responsibility of the University of Minnesota.

The automated logic of the REDCap database system will enable complete records. All data are by self report.
## 11 STATISTICAL CONSIDERATIONS

# 11.1 Study Hypotheses

We hypothesize that hydroxychloroquine is superior to placebo for preventing progression to COVID-19 disease among those who are asymptomatic.

We hypothesize that hydroxychloroquine is superior to placebo for preventing progression among those with symptomatic mild COVID19 disease preventing hospitalization/death.

# 11.2 Sample Size Considerations

Two cohorts of 1500 subjects each:

- 1) Asymptomatic persons exposed to COVID-19 disease (750 in placebo, 750 in intervention);
- 2) Symptomatic outpatient COVID-19 disease (750 in placebo, 750 in intervention).

Assuming 90% power, a two-sided alpha = 0.05 and loss to follow-up up to 20%, for each cohort the planned sample size is 750 participants per arm based on the following assumptions:

- 10% transmission rate from COVID-19 cases to close contacts
- For those with symptomatic illness the proportions at day 14 in the placebo group are 90%, 8% and 2%, respectively for illness without hospitalization, hospitalization with ICU stay or death, and hospitalization with an ICU stay or death.

The estimated transmission rates are uncertain. Table 1 below (for the asymptomatic cohort with exposure) shows that we are well powered to detect even a smaller (40%) relative reduction in the incidence of COVID 19 with 80% power for transmission rates of at least 10% with placebo. Table 2 (for the symptomatic group) shows that we are well powered to detect a common odds ratio of 0.6-0.75 under the assumption that the control proportions for illness without hospitalization, hospitalization without ICU stay or death and hospitalization with ICU stay or death are 90%, 8% and 2%, respectively.

**Table 1. Sample Size Table for Asymptomatic Participants** (Healthcare worker or household contact) With Exposure

| Estimated transmission rate with placebo | Estimated<br>transmission rate<br>with drug | Percent relative reduction in transmission rate | Sample size<br>(per arm) with<br>90% power | Sample size<br>(per arm) with<br>80% power |
|---|---|---|---|---|
| 10% | 5% | 50% | 621 | 474 |
| | 6% | 40% | 1014 | 771 |
| 12% | 6% | 50% | 509 | 389 |
| | 7.2% | 40% | 831 | 632 |
| 15% | 7.5% | 50% | 398 | 304 |
| | 9% | 40% | 648 | 493 |

**Table 2. Sample size table for participants with symptomatic disease**, assuming that the control proportions are 90% illness with no hospitalization, 8% hospitalization with no ICU stay or death and 2% hospitalization with ICU stay or death.

| Log Odds Ratio | Odds Ratio | Sample size (per<br>group) with 90%<br>power | Sample size (per<br>group) with 80%<br>power |
|---|---|---|---|
| 0.60 | 1.82 | 805 | 601 |
| 0.65 | 1.91 | 697 | 521 |
| 0.70 | 2.01 | 610 | 456 |
| 0.75 | 2.12 | 539 | 403 |

# 11.3 Planned Interim Analyses

A Lan-DeMets spending function analog of the O'Brien-Fleming boundaries will be provided at each DSMB report for the primary outcome for each cohort. The O'Brien-Fleming boundaries will be truncated at alpha = 0.001 (|Z| > 3.09). For each cohort, interim analyses are separately planned at 25%, 50% and 75% of trial enrollment.

As enrollment may be brisk, the timing of interim analyses may be altered at PI discretion based on that pace of enrollment. It may be possible that the trial is fully enrolled by the time day 14 outcomes are available for the first 25% enrolled. In this case, any further analyses would be related as to when to release interim results.

At the first DSMB review, the stopping boundary is unlikely to be crossed. The purpose of this early review will assess the trends for safety/efficacy and allow for the DSMB to determine the probable timing of further reviews based on the pace of enrollment.

Should a stopping boundary be crossed, we would recommend an analysis to determine whether the findings are consistent across secondary endpoints, such that a clear answer is achieved. Starting with the 2<sup>nd</sup> DSMB review (at approximately 50% enrollment) the DSMB will be given the conditional power for both cohorts under both the study design parameters and the current data. If the conditional power is less than 20% then trial discontinuation may be considered.

In the event of early halting due to efficacy of the intervention, the study will immediately convert to an open label observational cohort of hydroxychloroquine prescribed to all consented participants in the relevant cohort.

In the event of early halting due to futility of no effect, a protocol modification will be made to alter the intervention.

Based on the public health situation, the DSMB has the prerogative to alter the stopping rules.

#### Sample Size Re-estimation:

At time of ~50% enrollment, a sample size re-estimation should occur based on the disease transmission rate in the control group. The *a priori* assumption (based on limited data) is 10% transmission risk. The new sample size estimation will take into account the updated transmission rate with no treatment and will be powered to detect a 50% relative reduction in outcome.

# 11.4 Final Analysis Plan

Primary outcome analyses (intention to treat):

#### Asymptomatic Cohort Primary Analysis:

Those with asymptomatic exposure: Incidence of COVID 19 disease by day 14 will be assessed via Fisher's Exact Test.

#### **Symptomatic Cohort Primary Analysis:**

Those with symptomatic disease at study entry: For a summary metric of the change in symptom severity over 14 days, a longitudinal change over time repeated measures mixed-regression model will estimate the treatment effect by study arm. Subjects without symptoms are coded as a zero severity. Persons hospitalized or dead are coded as 10 severity.

Participants who become symptomatic with COVID19 on Day 1 before receiving the study medicine will be described with the symptomatic cohort.

#### Secondary Analyses:

For the asymptomatic with exposure cohort, the primary analysis (intention to treat) will be repeated for participants who received at least one dose of the study medicine.

- Secondary endpoints will be assessed via Fisher's Exact test and median (with interquartile ranges) as appropriate.
- Those with symptomatic disease at study entry: Proportional odds models will be used
  to assess the ordinal scale for disease severity at day 14 (illness without hospitalization,
  hospitalization without ICU stay or death).
- Severity of overall symptoms at Day 0, 1, 5, and 14 is recorded on a 0-10 visual analog scale. Severity of symptoms at Day 5 will be compared first as a categorical analysis (no symptoms vs. symptoms) via Fisher's Exact Chi Square.
  - Second among those with symptoms, the 0-10 visual analog scale severity data will be compared via independent two-sample t test. If data are non-normally distributed, then data will be compared via Mann-Whitney U by study arm.

A priori subgroup analyses will include assessment by:

- Confirmed SARS-CoV-2 disease or disease exposure
- Healthcare worker vs. Household contact
- Days from Exposure
- Decile of age
- Sex as a biological variable
- Censored subjects, who became symptomatic before receipt of the first dose of study medicine on D#1, will be separately analyzed and reported.

#### Handling of withdrawn subjects.

If there is a large lost to follow up / study discontinue rate, then the primary endpoint for the asymptomatic cohort would have a secondary analysis to assess incidence as a 3-category analysis of: i) no disease, ii) incident disease, or iii) unknown.

Similarly, the symptomatic cohort would add a fourth category of unknown.

Participants who stop taking the study medicine but who agree to be followed for 14 days will be assessed as intent-to-treat. On Day 14, we will ask for other medications or vitamins that were taken during the study period.

#### **Screened Persons**

Persons who are screened but not enrolled will be summarized in CONSORT diagrams and other descriptive summaries of their COVID-19 related information – with all data de-identified.

## 12 Source Documents and Access to Source Data

Source documents will include internet forms self-completed by participants directly entered into a RedCAP database.

This protocol is based on self-report.

This internet-based protocol is meant to enable a large number of participants to be recruited, quickly as well as maintain the safety of the research staff. In person visits, create a public health

Participants will be asked to provide consent to obtain medical records from their healthcare provider or public health official, if there is the need to verify outcomes – for SARS-CoV-2 test results or hospitalizations.

# 13 QUALITY CONTROL AND QUALITY ASSURANCE

Study medications will be commercially procured U.S. FDA-approved hydroxychloroquine or under ANDA #210959 following Good Manufacturing Practice.

## 14 ETHICS/PROTECTION OF HUMAN SUBJECTS

## 14.1 Ethical Standard

This study is to be conducted according to US and international standards of Good Clinical Practice (International Conference on Harmonization guidelines), Declaration of Helsinki, and International Ethical Guidelines for Biomedical Research Involving Human Subjects, applicable U.S. government regulations and institutional research policies and procedures. All investigators must have received human subject protection and GCP training prior to human subject involvement.

#### 14.2 Institutional Review Board

Prior to the initiation of the study, the protocol, all informed consent forms and the participant Information materials will be submitted to and approved by the single IRB of record. Likewise, any future amendments to the study protocol will be submitted and approved by the IRB before implementation. This protocol and any amendments will undergo review and approval by the Human Subjects Board at the University of Minnesota under DHHS Assurance FWA00000312.

## 14.3 Informed Consent Process

- Written informed consent will be obtained via an English-language, internet-based web
  form. If potential participants have questions, they may contact <a href="mailto:faq.covid19@gmail.com">faq.covid19@gmail.com</a>
  to reach a study staff member to answer their questions about research, either via email
  or a phone call.
- After completion of reading the form, participants will be assessed for comprehension, querying:
  - Concept of Randomization to hydroxychloroquine or vitamin placebo
  - Whether hydroxychloroquine is known to be effective in preventing disease
  - Duration of the study? (14 days)
  - Duration of taking the study medicine (5 days)
  - When follow up surveys will be sent (Days 1, 3, 5, 10 and 14)
  - If hydroxychloroquine can be shared? (No)

## 14.3.1 Informed Consent/Assent Process (in Case of a Minor)

Persons under 18 years of age are not eligible to participate. COVID19 has
negligible mortality in children <10 years, and rate of progression to symptomatic
disease may likely be different. Furthermore, pediatric dosing is weight based,
making remote administration more complicated with fixed dose 200mg tablets.</li>

## 14.4 Exclusion of Women, Minorities, and Children

 Persons under 18 years of age are not eligible to participate. COVID19 has 0% mortality in children and young adults.

 Non-English speaking adults are not eligible as the webpage and consents will only be available in English.

# 14.5 Subject Confidentiality

- Interaction will be via internet-based RedCAP ECRFs conforming to required U.S. privacy and server security standards.
- Clinical data will be entered into a study specific database by designated staff on a regular basis from completed electronic Case Record Forms (eCRF). Access to database will be given to authorized personnel only (members of the immediate study team). eCRF and trial documents will be kept in a secure database.
- Documentation, data and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party, without prior written approval of the participant except as necessary for monitoring by the IRB or public health authorities
- No participant identifying information will be disclosed in any publication or at any conference activities arising from the study.

# 14.6 Future Use of Stored Specimens

• No specimens are to be stored for future research.

## 15 DATA HANDLING AND RECORD KEEPING

## 15.1 Data Management Responsibilities

Investigators will maintain a REDCAP database of study records.

Survey forms will be self-completed by study participants.

# 15.2 Data Capture Methods

• Data will be obtained via internet-based REDCAP forms.

# 15.3 Types of Data

 Participants will be asked to provide data regarding COVID19 exposure timing and location. They will also be asked to provide ongoing symptom reports during the follow-up period.

## 15.4 Timing/Reports

- An enrollment progress report will be generated monthly
  - Participants Enrolled
  - o Participants on study
  - Participants completed the study
  - Lost to Follow Up
  - Cumulative COVID19 (pooled, both arms)
  - Cumulative Hospitalizations (pooled, both arms)
- A data safety monitoring board (DSMB) will review data after every 100 participants complete 14 days of follow-up.
- De-identified data will be shared with the research team members for analysis.

# 15.5 Study Records Retention

- No paper documents will be retained or stored.
- Digital records will be kept in a secure server setting.

## 15.6 Protocol Deviations

Protocol violations will be reported to the IRB of record.

## 16 Publication Policy

Publication will be expeditiously made with a full, de-identified data made available.

# 17 LITERATURE REFERENCES

Report of the WHO-China Joint Mission on Coronavirus Disease 2019 (COVID-19).
 2020. Available at: <a href="https://www.who.int/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf">https://www.who.int/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf</a>

- 2. Wang M, Cao R, Zhang L, et al. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. *Cell Res* 2020; 30: 269-71.
- 3. Vincent MJ, Bergeron E, Benjannet S, et al. Chloroquine is a potent inhibitor of SARS coronavirus infection and spread. *Virol J* 2005; 2: 69.
- 4. Cong Y, Hart BJ, Gross R, et al. MERS-CoV pathogenesis and antiviral efficacy of licensed drugs in human monocyte-derived antigen-presenting cells. *PLoS One* 2018; 13: e0194868.
- 5. Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In vitro antiviral activity and projection of optimized dosing design of hydroxychloroquine for the treatment of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). *Clin Infect Dis.* 202. *In Press.* doi: 10.1093/cid/ciaa237.
- 6. Burke RM, Midgley CM, Dratch A, Fenstersheib M, Haupt T, Holshue M, Ghinai I, Jarashow MC, Lo J, McPherson TD, Rudman S, Scott S, Hall AJ, Fry AM, Rolfes MA. Active monitoring of persons exposed to patients with confirmed covid-19 United States, January-February 2020. MMWR Morb Mortal Wkly Rep. 2020;69:245-6.
- 7. Lim HS, Im JS, Cho JY, Bae KS, Klein TA, Yeom JS, Kim TS, Choi JS, Jang IJ, Park JW. Pharmacokinetics of hydroxychloroquine and its clinical implications in chemoprophylaxis against malaria caused by Plasmodium vivax. *Antimicrob Agents Chemother*. 2009;53:1468-75. PMCID: 2663072.
- 8. Carmichael SJ, Charles B, Tett SE. Population pharmacokinetics of hydroxychloroquine in patients with rheumatoid arthritis. *Therapeutic Drug Monitoring*. 2003;25:671-81.
- Haeusler IL, Chan XHS, Guerin PJ, White NJ. The arrhythmogenic cardiotoxicity of the quinoline and structurally related antimalarial drugs: A systematic review. *BMC Med*. 2018;16:200. PMCID: PMC6220451.

## **SUPPLEMENTS / APPENDICES**

#### **APPENDIX A: SCHEDULE OF EVENTS**

#### **Overview of Procedures**



Participants with ongoing SAE / hospitalization at day 14 will be followed until hospital discharge or up to day 90 for final resolution.

- 1. Report of the WHO-China Joint Mission on Coronavirus Disease 2019 (COVID-19). **2020**.
- 2. Wang M, Cao R, Zhang L, et al. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. *Cell Res* **2020**; 30: 269-71.
- 3. Vincent MJ, Bergeron E, Benjannet S, et al. Chloroquine is a potent inhibitor of SARS coronavirus infection and spread. *Virol J* **2005**; 2: 69.
- 4. Cong Y, Hart BJ, Gross R, et al. MERS-CoV pathogenesis and antiviral efficacy of licensed drugs in human monocyte-derived antigen-presenting cells. *PLoS One* **2018**; 13: e0194868.
- 5. Yao X, Ye F, Zhang M, et al. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). *Clin Infect Dis* **2020**; *In Press*.
- 6. Pastick KA, Okafor EC, Wang F, et al. Review: Hydroxychloroquine and Chloroquine for Treatment of SARS-CoV-2 (COVID-19). *Open Forum Infectious Diseases* **2020**; ofaa130.
- 7. Chen J, Liu D, Liu L, et al. A pilot study of hydroxychloroquine in treatment of patients with common coronavirus disease-19 (COVID-19). *Journal of Zhejiang University* **2020**.
- 8. Gautret P, Lagier JC, Parola P, et al. Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. *Int J Antimicrob Agents* **2020**; 105949.
- 9. Chen Z, Hu J, Zhang Z, et al. Efficacy of hydroxychloroquine in patients with COVID-19: results of a randomized clinical trial. *medRxiv* **2020**.
- 10. Molina JM, Delaugerre C, Goff JL, et al. No Evidence of Rapid Antiviral Clearance or Clinical Benefit with the Combination of Hydroxychloroquine and Azithromycin in Patients with Severe COVID-19 Infection. *Médecine et Maladies Infectieuses* **2020**.
- 11. Gautret P, Lagier JC, Parola P, et al. Clinical and microbiological effect of a combination of hydroxychloroquine and azithromycin in 80 COVID-19 patients with at least a six-day follow up: A pilot observational study. *Travel Med Infect Dis* **2020**; 101663.
- 12. Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. *Biosci Trends* **2020**; 14: 72-3.
- 13. Burke RM, Midgley CM, Dratch A, et al. Active Monitoring of Persons Exposed to Patients with Confirmed COVID-19 United States, January-February 2020. *MMWR Morb Mortal Wkly Rep* **2020**; 69: 245-6.
- 14. Haeusler IL, Chan XHS, Guerin PJ, White NJ. The arrhythmogenic cardiotoxicity of the quinoline and structurally related antimalarial drugs: a systematic review. *BMC Med* **2018**; 16: 200.
- 15. Lim HS, Im JS, Cho JY, et al. Pharmacokinetics of hydroxychloroquine and its clinical implications in chemoprophylaxis against malaria caused by Plasmodium vivax. *Antimicrob Agents Chemother* **2009**; 53: 1468-75.
- 16. Carmichael SJ, Charles B, Tett SE. Population Pharmacokinetics of Hydroxychloroquine in Patients With Rheumatoid Arthritis. *Therapeutic Drug Monitoring* **2003**; 25: 671-81.

# Post-exposure Prophylaxis or Preemptive Therapy for SARS-Coronavirus-2: A Pragmatic Randomized Clinical Trial

Statistical Analysis Plan
06 May 2020

| Protocol Version, Date | Primary Endpoint |
|--------------------------------------|-----------------------|
| Protocol Version 1.0, March 17, 2020 | Incidence of COVID19* |
| Protocol Version 2.0; March 20, 2020 | Incidence of COVID19 |
| Protocol Version 2.1, March 26, 2020 | Incidence of COVID19 |
| Protocol Version 2.2; March 27, 2020 | Incidence of COVID19 |
| Protocol Version 2.3, April 24, 2020 | Incidence of COVID19 |

<sup>\*</sup> Incidence of COVID19 disease, defined on March 17 and thereafter as: "The primary analysis will use PCR+ confirmed disease. However if the absence of sufficient testing supplies continues then outpatients will not be offered SARS-CoV-2 testing unless they are sick enough to be hospitalized. In that case an alternate a priori planned analysis will define incident COVID19 disease as a composite of SARS-CoV-2 PCR+ confirmed result OR symptomatic disease (i.e. possible) COVID-19 in those without testing."

## I. Prophylaxis study primary outcome

- a. The primary outcome will be presented for the treatment and control groups as proportions, and compared with Fisher's Exact tests.
- b. The primary outcome will be presented for subgroups formed by contact type (household contact and healthcare workers), age groups (18-35, 36-50 and > 50), sex, and days from exposure. These are apriori subgroups defined in the Version 1.0 of the protocol.
- c. Participants who are randomized into the prevention trial, but who become symptomatic on Day 1 before receiving the study medicine will be censored from the prevention cohort and analyzed with the companion treatment cohort.
- d. The primary outcome will be presented by subgroups formed by COVID test results (confirmed positive vs. other), age groups (18-35, 36-50, > 50), sex, and days from exposure onset to entry. These are apriori subgroups defined in the Version 1.0 of the protocol.
- e. Medication adherence is captured on study day 5. Another subgroup of interest is comparing the treatment groups for change in symptom severity score after day 5 by adherence reported at day 5 (<= 75% versus > 75%).

## II. Secondary outcomes

- a. Secondary outcomes for incidence will be presented as proportions and compared between the treatment groups with Fisher's Exact tests.
- b. Symptom severity scores were recorded with the online participant surveys at days 3, 5, 10 and 14 only for those who responded "yes" to "Any symptoms experienced".

i. Visual analog scale (0-10) for "overall symptom severity" is collected via a digital slider bar, which is marked with "0 = no symptoms"; 5 (placed in the middle); and "10 = severe symptoms"



- ii. For those who responded "no" to "Any symptoms experienced" the symptom severity score for that visit is assigned as zero.
- iii. For those hospitalized or with deaths, their symptom severity was scored as 10 if they did not respond to the visit survey.
- iv. Analysis is by Kruskall Wallis tests among those with symptoms at day 14.

## Clarifications (24 May 2020):

- Participants with missing outcome data are still included in the denominator, as the trial is performed as an intent to treat analysis.
- Sensitivity analyses were performed excluding participants with missing data from the denominator as well as including participants with missing data as events.